CLINICAL TRIAL: NCT05688891
Title: The Effect of Virtual Reality and Music on Pain, Anxiety and Pain Anxiety in Burn Patient Care
Brief Title: Burn Patient Care, Virtual Reality, Music, Pain, Anxiety and Pain Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Collaborators: Prof. Dr. SEHER DENİZ ÖZTEKİN (Unknown)
Responsible Party: Principal Investigator, RABİA GÖRÜCÜ, research assistant, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022/514/221/7
Record Dates: First submitted 2023-01-09; First posted 2023-01-18 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2023-01

CONDITIONS: PAIN; ANXIETY; PAIN ANXIETY
Keywords: Burn care; Pain; Anxiety; Pain anxiety; Nursing
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: prospective randomized controlled clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual reality (Experimental): Before the procedure, "Visual Analogue Scale-VAS", "Spielberger State and Trait Anxiety Inventory", "Burn-Specific Pain Anxiety Scale" were filled in.5 minutes before the burn dressing procedure, virtual reality glasses were put on the patient's head by the researcher and a 360° VR video with submarine and nature content pre-loaded on the glasses was opened.
  Video monitoring with Virtual Reality continued throughout the entire dressing.This procedure was performed during 2 consecutive dressing changes. A 1-week period was given between 2 dressings.After the procedure, the scales were filled again.
  Interventions: Other: Virtual reality
- Music (Experimental): 5 minutes before the burn dressing procedure, the patient was asked about the type of music he preferred in the introductory patient information form. Then, the patient was started to listen after putting on headphones and adjusting the volume. The patient was asked to keep his eyes closed while listening to music. Music listening was continued throughout the entire dressing.This procedure was performed during 2 dressing changes in accordance with clinical treatment and protocols.
  A 1-week period was given between 2 dressings.After the procedure, the scales were filled again.
  Interventions: Other: Music
- Control (No Intervention): During the burn dressing procedure, no intervention method was used, and routine treatment and care interventions were continued.This procedure was performed during 2 dressing changes in accordance with clinical treatment and protocols.
  A 1-week period was given between 2 dressings.

INTERVENTIONS:
Other: Virtual reality — 5 minutes before the burn dressing procedure, virtual reality glasses were put on the patient's head by the researcher and a 360° VR video with submarine and nature content pre-loaded on the glasses was opened.
  Audio and video settings were made and started to be watched. Video monitoring with Virtual Reality continued throughout the entire dressing. This procedure was performed during 2 consecutive dressing changes. A 1-week period was given between 2 dressings.
  Arms: Virtual reality
Other: Music — 5 minutes before the burn dressing procedure, the patient was asked about the type of music he preferred in the introductory patient information form. Then, the patient was started to listen after putting on headphones and adjusting the volume. The patient was asked to keep his eyes closed while listening to music. Music listening was continued throughout the entire dressing.
  After the process was finished, the music was turned off and the headphones were removed.
  This procedure was performed during 2 dressing changes in accordance with clinical treatment and protocols.
  A 1-week period was given between 2 dressings.
  Arms: Music

SUMMARY:
Different non-pharmacological methods such as virtual reality glasses and music can be applied by nurses within the scope of care interventions for the management of pain and anxiety in burn patients during dressing changes and debridement.

In this study, it was aimed to determine the effect of virtual reality and music on pain, anxiety and pain anxiety in burn patient care.

DETAILED DESCRIPTION:
Wound debridement, wound care, surgical interventions and other invasive procedures applied during burn treatment cause the patient to feel pain, and the repeated pain process creates anxiety in the patient.

In the studies in the literature, it is stated that anxiety and pain are closely related, pain affects the level of anxiety and anxiety affects the severity of pain.

The role of nurses in the burn team is very important in the management of pain and anxiety in the treatment of burns, which have both physiological and psychological effects.

The most important responsibility of the nurse in burn patient care is continuous and individualized pain diagnosis and management.

Different non-pharmacological methods such as virtual reality glasses and music can be applied by nurses within the scope of care interventions for the management of pain and anxiety.

Music is widely used to reduce pain and anxiety in burn patients during dressing changes and debridement.

Virtual reality (VR) glasses, which facilitate daydreaming and daydreaming, are another method used to reduce pain and anxiety. With the development of technology, the use of virtual reality glasses by nurses as a method of distraction, especially in burn patients, is increasing.

In this study, it was aimed to determine the effect of virtual reality and music on pain, anxiety and pain anxiety in burn patient care.

The sample group was selected in accordance with the research criteria from the individuals in the population who were given permission to participate in the research after the purpose of the research was explained.

Within the scope of the planned study, the sample size to be used in determining the effect of virtual reality and music on pain, anxiety and pain anxiety in burn patient care, effect size d= 0.485 (effect size), α=0.05 ( margin of error), 1-β With the help of the G-power (version 3.1) package program, a total of 120 people (at least 40 people in each group) were calculated, as =0.80 (power).

A list was created for 120 patients who met the inclusion criteria in the study and distributed to the experimental and control groups using a computerized randomization program.

ELIGIBILITY:
Inclusion Criteria:

* be between the ages of 18-65,
* Ability to read, write and speak Turkish,
* Not participating in another clinical trial at the same time,
* Not having any problems that prevent cognitive, affective and verbal communication,
* Having a patient group with a burnt total body area (TBSA) of less than 15%,
* 2nd degree and 3rd degree patient group in the granulation stage,
* No burns on the head, ears and face,
* Being a patient group with daily dressing changes and dressing frequency of 1-15,
* Absence of complaints such as respiratory problems that would prevent him from participating in the study,
* Absence of vision and hearing problems.

Exclusion Criteria:

* Pain intensity is between 8-10 points,
* Being under the influence of pharmacological or non-pharmacological intervention that will affect the pain,
* Being a first degree patient group,
* Having neurological, psychological and psychiatric diseases,
* Burns on the head, ears and face,
* Having vision and hearing problems,
* Applying sedation to the patient during the dressing,
* Stop watching VR glasses during dressing,
* Stop listening to music during dressing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2023-01-14 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
Pain evaluated using Visual Analog Scale | Change from baseline (before implementation) and 2th week of practice
  Visual Analog Scale (VAS) is the most frequently used and simplest to use scale. In the scale with numbers between 0-10, "0" defines painlessness and "10" defines the most severe pain.
  In order to define the numerical value of the patient's pain/anxiety severity, the patient is asked to mark the ruler consisting of a 10 cm line, and the patient's pain severity score is determined as a result of the measurement.
  The scale consists of five parts. Each of the sections is in the range of 2 points. '0' points - no pain, '1-2 points, very mild pain', '3-4 points, mild pain', '5-6 points, moderate pain', '7-8 points, severe pain' means '9-10 points, excruciating pain'.
Anxiety evaluated using The State Anxiety Inventory | Change from baseline (before implementation) and 2th week of practice
  It is a self-assessment scale consisting of twenty items developed by Spielberger et al. (1970) to determine state anxiety levels. The Turkish validity and reliability study of this scale was performed by Öner and LeCompte (1977), and the internal consistency (Cronbach's Alpha) coefficients were found to be between 0.83 and 0.92 for the state anxiety scale (Öner & LeCompte, 1998). Higher total scores on the scale indicate a high level of state anxiety.
  The response options collected in four classes in the state anxiety scale are (1) Not at all, (2) Somewhat, (3) A lot, and (4) Completely. There are ten reversed statements in the state anxiety scale. These are items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20.
  The scores obtained in the scale theoretically vary between 20 and 80. A large score indicates a high level of anxiety, and a small score indicates a low level of anxiety.
Pain Anxiety evaluated using The Burn Specific Pain Anxiety Scale (BSPAS) | Change from baseline (before implementation) and 2th week of practice
  The Burn Specific Pain Anxiety Scale (BSPAS) is another tool which evaluates pain related anxiety in burn patients. For each question in this scale, 0 "never" and 10 "worst possible" are accepted. The scale total score is calculated by summing the scores of all items and the lowest score is 0 and the highest score is 80. The higher the total score, the higher the anxiety experienced by the patient about painful procedures while in the hospital.

SECONDARY OUTCOMES:
Anxiety evaluated using The Trait Anxiety Inventory | State from baseline (before implementation)
  In the trait anxiety scale, the number of reversed statements is seven and these make up the items 21, 26, 27, 30, 33, 36 and 39. On the trait anxiety scale, reversed statements the number of statements is seven and these make up Articles 21, 26, 27, 30, 33, 36 and 39.
  The scores obtained from both scales theoretically vary between 20 and 80. A large score indicates a high level of anxiety, and a small score indicates a low level of anxiety. The same is true when interpreting scores in percentile order. That is, the low percentile rank (1, 5, 10) indicates less anxiety. The average score level determined in the applications varies between 36 and 41.

CONTACTS AND LOCATIONS:
Locations (1):
- Turkey, Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No